CLINICAL TRIAL: NCT01606007
Title: A Multicenter, Randomized, Double-Blind, Active Controlled, Parallel Group, Phase 3 Trial to Evaluate the Safety and Efficacy of Add-On Therapy With Saxagliptin and Dapagliflozin Added to Metformin Compared to Add-On Therapy With Saxagliptin in Combination With Metformin or Dapagliflozin in Combination With Metformin in Subjects With Type 2 Diabetes Who Have Inadequate Glycemic Control on Metformin Alone.
Brief Title: Safety and Efficacy of Combination Saxagliptin & Dapagliflozin Added to Metformin to Treat Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CV181-169; 2012-000679-18 (EudraCT Number)
Record Dates: First submitted 2012-05-23; First posted 2012-05-25 (Estimated); Results first posted 2015-10-20 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-03

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — saxagliptin; Metformin; dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1: Saxagliptin+Metformin XR+Placebo (Active Comparator)
  Interventions: Drug: Saxagliptin; Drug: Metformin XR; Drug: Placebo matching with Dapagliflozin
- Arm 2: Dapagliflozin+Metformin XR+Placebo (Active Comparator)
  Interventions: Drug: Metformin XR; Drug: Dapagliflozin; Drug: Placebo matching with Saxagliptin
- Arm 3: Saxagliptin+Dapagliflozin+Metformin XR (Experimental)
  Interventions: Drug: Saxagliptin; Drug: Metformin XR; Drug: Dapagliflozin

INTERVENTIONS:
Drug: Saxagliptin — Tablets, Oral, 5mg , Once daily, 24 weeks
  Other Names: Onglyza
  Arms: Arm 1: Saxagliptin+Metformin XR+Placebo; Arm 3: Saxagliptin+Dapagliflozin+Metformin XR
Drug: Metformin XR — Tablets, Oral, ≥ 1500mg/≤ 2000mg, Once daily, 24 weeks
  Other Names: Glucophage XR
Drug: Dapagliflozin — Tablets, Oral, 10mg , Once daily, 24 weeks
  Other Names: BMS-512148
  Arms: Arm 2: Dapagliflozin+Metformin XR+Placebo; Arm 3: Saxagliptin+Dapagliflozin+Metformin XR
Drug: Placebo matching with Dapagliflozin — Tablets, Oral, 0mg, Once daily, 24 weeks
  Arms: Arm 1: Saxagliptin+Metformin XR+Placebo
Drug: Placebo matching with Saxagliptin — Tablets, Oral, 0mg, Once daily, 24 weeks
  Arms: Arm 2: Dapagliflozin+Metformin XR+Placebo

SUMMARY:
The purpose of this study is to learn if a combination of BMS-477118 (Saxagliptin) and BMS -512148 (Dapagliflozin) added to Metformin can improve (decrease) Glycosylated Hemoglobin (Hemoglobin A1c) in patients with type 2 diabetes after 24 weeks of treatment. The safety of this treatment will also be studied.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with Type 2 diabetes mellitus (T2DM) with HbA1c ≥ 8.0% and ≤ 12.0%
* Stable metformin therapy dose of ≥ 1500mg for at least 8 weeks prior to screening
* Body mass index (BMI) ≤ 45.0kg/m2

Exclusion Criteria:

* Estimated glomerular filtration rate (eGFR) < 60mL/min/1,73m2 and Serum Creatinine (Scr) ≥ 1.5 mg/dL in males or ≥ 1.4 mg/dL in females
* Uncontrolled hypertension Systolic Blood Pressure (SBP) ≥ 160mmHg and/or Diastolic Blood Pressure (DBP) ≥ 100mmHg
* Hepatic disease
* Cardiovascular disease within 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1282 (Actual)
Dates: Start 2012-07; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (129):
- United States (80):
  - Central Alabama Research, Birmingham, Alabama
  - Central Alabama Research, Homewood, Alabama
  - Terence T. Hart, Md, Muscle Shoals, Alabama
  - International Institute Of Clinical Research, Ozark, Alabama
  - Clinical Research Advantage, Mesa, Arizona
  - Elite Clinical Studies, Llc, Phoenix, Arizona
  - Genova Clinical Research, Tucson, Arizona
  - Medical Investigations, Inc., Little Rock, Arkansas
  - Aureus Research, Inc., Little Rock, Arkansas
  - Southland Clinical Research Center, Inc., Fountain Valley, California
  - Torrance Clinical Research, Lomita, California
  - National Research Inst, Los Angeles, California
  - Providence Clinical Research, North Hollywood, California
  - Diabetes Medical Center Of California, Northridge, California
  - Mehrdad Kevin Ariani Md, Inc., Northridge, California
  - Lucita M. Cruz,Md.,Inc., Norwalk, California
  - Center For Clinical Trials, Llc., Paramount, California
  - Center For Clinical Trials Of Sacramento, Inc., Sacramento, California
  - Trinitas Research, Inc, San Jose, California
  - Orange County Research Center, Tustin, California
  - Clinical Research Advantage, Colorado Springs, Colorado
  - Infocus Clinical Research, Denver, Colorado
  - Lynn Institute Of Denver, Denver, Colorado
  - Southeast Clinical Research, Llc, Chiefland, Florida
  - Clinical Therapeutics Corporation, Coral Gables, Florida
  - Southeast Clinical Research, Llc, Jacksonville, Florida
  - Fpa Clinical Research, Kissimmee, Florida
  - Clinical Research Of Miami, Inc., Miami, Florida
  - Advanced Pharma Cr, Llc, Miami, Florida
  - Newphase Clinical Trials, Inc., Miami Beach, Florida
  - Omega Research Consultants, Llc, Orlando, Florida
  - Palm Harbor Medical Associates, Palm Harbor, Florida
  - Andres Patron, Do Pa, Pembroke Pines, Florida
  - Endocrine Research Solutions, Inc., Roswell, Georgia
  - Cedar Crosse Research Center, Chicago, Illinois
  - Deerbrook Medical Associates, Vernon Hills, Illinois
  - Clinical Research Advantage, Council Bluffs, Iowa
  - Horizon Research Group Of Opelousas, Llc, Eunice, Louisiana
  - Associated Internal Medicine Specialists, Battle Creek, Michigan
  - Harris And Associates, P.C., Detroit, Michigan
  - Patterson Medical Clinic, Florissant, Missouri
  - Bellevue Family Practice, Bellevue, Nebraska
  - Clinical Research Advantage, Elkhorn, Nebraska
  - Clinical Research Advantage, Fremont, Nebraska
  - Clinical Research Advantage, Omaha, Nebraska
  - South Jersey Medical Associates, P.A., Blackwood, New Jersey
  - Central Jersey Health And Medical Research, Elizabeth, New Jersey
  - Southgate Medical Group, West Seneca, New York
  - Metrolina Internal Medicine, Charlotte, North Carolina
  - Triad Clinical Trials, Llc, Greensboro, North Carolina
  - Diabetes & Endocrinology Consultants, Morehead City, North Carolina
  - Pmg Research Of Winston-Salem, Llc, Winston-Salem, North Carolina
  - Daystar Clinical Resarch, Inc., Akron, Ohio
  - Sterling Research Grp, Ltd., Cincinnati, Ohio
  - Rapid Medical Research, Inc., Cleveland, Ohio
  - Primed Clinical Research, Dayton, Ohio
  - Physicians Research, Inc., Zanesville, Ohio
  - Lynn Institute Of Norman, Norman, Oklahoma
  - Willamette Valley Clinical Studies, Eugene, Oregon
  - Oregon Clinical Research, Portland, Oregon
  - Heritage Valley Medical Group, Beaver, Pennsylvania
  - Wellmon Family Practice, Shippensburg, Pennsylvania
  - Tlm Medical Services, Columbia, South Carolina
  - Palmetto Clinical Trial Services Llc, Fountain Inn, South Carolina
  - Holston Medical Group, Bristol, Tennessee
  - Holston Medical Group, Kingsport, Tennessee
  - Pmg Research Of Knoxville, Knoxville, Tennessee
  - Arlington Family Research Center, Inc., Arlington, Texas
  - Padre Coast Clinical Research, Corpus Christi, Texas
  - Dallas Diabetes & Endocrine Center, Dallas, Texas
  - Excel Clinical Research, Llc, Houston, Texas
  - North Hills Medical Research, Inc., North Richland Hills, Texas
  - Med-Olam Clinical Research, Pasadena, Texas
  - Sam Clinical Research Center, San Antoinio, Texas
  - Covenant Clinical Research, Pa, San Antonio, Texas
  - Hillcrest Family Health Center, Waco, Texas
  - Val R. Hansen, M.D., Bountiful, Utah
  - Highland Clinical Research, Salt Lake City, Utah
  - Southwestern Vermont Med Cntr, Bennington, Vermont
  - Hampton Roads Center For Clinical Research, Inc., Suffolk, Virginia
- Canada (8):
  - Local Institution, Coquitlam, British Columbia
  - Local Institution, Winnipeg, Manitoba
  - Local Institution, Brampton, Ontario
  - Local Institution, Smiths Falls, Ontario
  - Local Institution, Toronto, Ontario
  - Local Institution, Granby, Quebec
  - Local Institution, Québec, Quebec
  - Local Institution, Saskatoon, Saskatchewan
- Mexico (7):
  - Local Institution, Aguascalientes, Aguascalientes
  - Local Institution, Chihuahua City, Chihuahua
  - Local Institution, Durango, Durango
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, Cuautla, Morelos
  - Local Institution, Monterrey, Nuevo León
  - Local Institution, Mérida, Yucatán
- Poland (8):
  - Local Institution, Gdansk
  - Local Institution, Katowice
  - Local Institution, Krakow
  - Local Institution, Lodz
  - Local Institution, Opole
  - Local Institution, Poznan
  - Local Institution, Puławy
  - Local Institution, Warsaw
- Puerto Rico (5):
  - Local Institution, Cidra
  - Local Institution, Manatí
  - Local Institution, Ponce
  - Local Institution, San Juan
  - Local Institution, Villa Fontana
- Romania (6):
  - Local Institution, Galati, Galați County
  - Local Institution, Ploieşti, Prahova
  - Local Institution, Timișoara, Timiș County
  - Local Institution, Bucharest
  - Local Institution, Cluj Napoca Cluj
  - Local Institution, Craiova
- South Africa (10):
  - Local Institution, Soweto, Gauteng
  - Local Institution, Gauteng, Johannesburg
  - Local Institution, Johannesburg, Johannesburg
  - Local Institution, Durban, KwaZulu-Natal
  - Local Institution, Cape Town, Western Cape
  - Local Institution, Goodwood, Western Cape
  - Local Institution, Paarl, Western Cape
  - Local Institution, Rondebosch, Western Cape
  - Local Institution, Somerset West, Western Cape
  - Local Institution, Johannesburg
- South Korea (5):
  - Local Institution, Bucheon-si, Gyeonggi-do
  - Local Institution, Sungnam-si, Gyeonggi-do
  - Local Institution, Daegu
  - Local Institution, Incheon
  - Local Institution, Seoul

REFERENCES:
- [Result] Rosenstock J, Hansen L, Zee P, Li Y, Cook W, Hirshberg B, Iqbal N. Dual add-on therapy in type 2 diabetes poorly controlled with metformin monotherapy: a randomized double-blind trial of saxagliptin plus dapagliflozin addition versus single addition of saxagliptin or dapagliflozin to metformin. Diabetes Care. 2015 Mar;38(3):376-83. doi: 10.2337/dc14-1142. Epub 2014 Oct 28. PMID 25352655
- [Derived] Bailey CJ, Del Prato S, Wei C, Reyner D, Saraiva G. Durability of glycaemic control with dapagliflozin, an SGLT2 inhibitor, compared with saxagliptin, a DPP4 inhibitor, in patients with inadequately controlled type 2 diabetes. Diabetes Obes Metab. 2019 Nov;21(11):2564-2569. doi: 10.1111/dom.13841. Epub 2019 Aug 26. PMID 31364269
- [Derived] Rosenstock J, Mathieu C, Chen H, Garcia-Sanchez R, Saraiva GL. Dapagliflozin versus saxagliptin as add-on therapy in patients with type 2 diabetes inadequately controlled with metformin. Arch Endocrinol Metab. 2018 Aug;62(4):424-430. doi: 10.20945/2359-3997000000056. PMID 30304106
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx
- See also: CV_181169_Protocol_Redacted — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3665&filename=CV_181169_Protocol_Redacted.pdf
- See also: CV181169_Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3665&filename=CV181169_Synopsis.pdf

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 1282 participants enrolled subjects, 534 eligible subjects entered the randomized, double-blind treatment period.
  Of 534 randomized and treated subjects, 490 subjects completed the study.
Groups:
- Arm 1: Saxagliptin+Metformin XR+Placebo: Drug: Saxagliptin Tablets, Oral, 5mg , Once daily, 24 weeks Other Names: Onglyza Drug: Metformin XR Tablets, Oral, ≥ 1500mg/≤ 2000mg, Once daily, 24 weeks Other Names: Glucophage XR Drug: Placebo matching with Dapagliflozin Tablets, Oral, 0mg, Once daily, 24 weeks
- Arm 2: Dapagliflozin+Metformin XR+Placebo: Drug: Metformin XR Tablets, Oral, ≥ 1500mg/≤ 2000mg, Once daily, 24 weeks Other Names: Glucophage XR Drug: Dapagliflozin Tablets, Oral, 10mg , Once daily, 24 weeks Other Names: BMS512148 Drug: Placebo matching with Saxagliptin Tablets, Oral, 0mg, Once daily, 24 weeks
- Arm 3: Saxagliptin+Dapagliflozin+Metformin XR: Drug: Saxagliptin Tablets, Oral, 5mg , Once daily, 24 weeks Other Names: Onglyza Drug: Metformin XR Tablets, Oral, ≥ 1500mg/≤ 2000mg, Once daily, 24 weeks Other Names: Glucophage XR Drug: Dapagliflozin Tablets, Oral, 10mg , Once daily, 24 weeks Other Names: BMS512148
Period: Overall Study
Arm/Group | Arm 1: Saxagliptin+Metformin XR+Placebo | Arm 2: Dapagliflozin+Metformin XR+Placebo | Arm 3: Saxagliptin+Dapagliflozin+Metformin XR
Started | 176 | 179 | 179
Completed | 161 | 160 | 169
Not Completed | 15 | 19 | 10
Not completed — Reason 'Other' in the protocol | 0 | 1 | 1
Not completed — Pregnancy | 0 | 1 | 1
Not completed — Withdrawal by Subject | 8 | 6 | 1
Not completed — Adverse Event | 0 | 1 | 1
Not completed — discontinue study treatment | 0 | 2 | 1
Not completed — Lost to Follow-up | 6 | 8 | 5
Not completed — Poor/Non-compliance | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Saxagliptin+Metformin XR+Placebo | Arm 2: Dapagliflozin+Metformin XR+Placebo | Arm 3: Saxagliptin+Dapagliflozin+Metformin XR | Total
Number analyzed (Participants) | 176 | 179 | 179 | 534
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.6 (9.6) | 53.5 (9.7) | 53.4 (9.8) | 53.8 (9.7)
Age, Customized [Number; unit: participants]
  <65 years | 148 | 158 | 160 | 466
  >=65 years | 28 | 21 | 19 | 68
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 90 | 94 | 266
  Male | 94 | 89 | 85 | 268
Race/Ethnicity, Customized [Number; unit: participants]
  White | 121 | 131 | 120 | 372
  Black african/american | 22 | 16 | 22 | 60
  Asian | 11 | 10 | 12 | 33
  Other | 22 | 22 | 25 | 69
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 31.8 (5.142) | 31.46 (5.321) | 31.76 (4.787) | 31.67 (5.080)
T2DM duration [Mean (Standard Deviation); unit: years] | 8.2 (5.52) | 7.4 (5.40) | 7.1 (5.04) | 7.6 (5.33)
HbA1c [Mean (Standard Deviation); unit: %] | 9.03 (1.05) | 8.87 (1.16) | 8.92 (1.18) | 8.94 (1.13)

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Mean Change From Baseline in Hemoglobin A1C (HbA1c) at Week 24
Description: HbA1c was measured as percent of hemoglobin by a central laboratory. Baseline was defined as the last assessment on or prior to the date of the first dose of the double-blind study medication. HbA1c measurements were obtained at Week 24 in the double-blind period, including observations prior to rescue.
Time Frame: Baseline (Week 0) and at Week 24
Population: All randomized participants who received study medication and had nonmissing HbA1c values at baseline and Week 24
Measure: Mean (95% Confidence Interval); unit: % HbA1c
Arm/Group | Arm 1: Saxagliptin+Metformin XR+Placebo | Arm 2: Dapagliflozin+Metformin XR+Placebo | Arm 3: Saxagliptin+Dapagliflozin+Metformin XR
Number analyzed (Participants) | 143 | 151 | 158
% HbA1c | -0.88 [-1.03 to -0.72] | -1.20 [-1.35 to -1.04] | -1.47 [-1.62 to -1.31]
Statistical Analysis 1: Comparison: Arm 1: Saxagliptin+Metformin XR+Placebo vs Arm 3: Saxagliptin+Dapagliflozin+Metformin XR; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Primary endpoint was tested at alpha=0.05; significance was claimed only if Saxagliptin+Dapagliflozin+Metformin was superior to both Saxagliptin+Metformin and Dapagliflozin+Metformin; Mean Difference (Final Values) = -0.59, 95% CI 2-sided [-0.81 to -0.37], Standard Error of Mean 0.1112
Statistical Analysis 2: Comparison: Arm 2: Dapagliflozin+Metformin XR+Placebo vs Arm 3: Saxagliptin+Dapagliflozin+Metformin XR; Test type: Superiority or Other; p = 0.0166, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.27, 95% CI 2-sided [-0.48 to -0.05], Standard Error of Mean 0.1108

2. Secondary Outcome: Adjusted Mean Change From Baseline in 2-hour Post Prandial Glucose (PPG) From a Liquid Meal Tolerance Test (MTT) at Week 24 (Last Observation Carried Forward [LOCF])
Description: Baseline was defined as the last assessment on or prior to the date of the first dose of the double-blind study medication. PPG measurements were obtained at week 24 in the doubleblind period, including observations prior to rescue.
Time Frame: Baseline (Week 0) and at Week 24
Population: All randomized participants who received study medication and had nonmissing PPG values at baseline and Week 24 (LOCF)
Measure: Mean (95% Confidence Interval); unit: MG/DL PPG
Arm/Group | Arm 1: Saxagliptin+Metformin XR+Placebo | Arm 2: Dapagliflozin+Metformin XR+Placebo | Arm 3: Saxagliptin+Dapagliflozin+Metformin XR
Number analyzed (Participants) | 147 | 144 | 154
MG/DL PPG | -35.6 (3.510) [-42.5 to -28.7] | -70.4 (3.538) [-77.4 to -63.5] | -79.6 (3.426) [-86.3 to -72.8]
Statistical Analysis 1: Comparison: Arm 1: Saxagliptin+Metformin XR+Placebo vs Arm 3: Saxagliptin+Dapagliflozin+Metformin XR; LOCF; Test type: Superiority or Other; p < 0.0001, ANCOVA — Each secondary endpoint was tested at alpha=0.05; significance was claimed only if Saxagliptin+Dapagliflozin+Metformin was superior to both Saxagliptin+Metformin and Dapagliflozin+Metformin; Mean Difference (Final Values) = -44.0, 95% CI 2-sided [-53.7 to -34.3], Standard Error of Mean 4.914
Statistical Analysis 2: Comparison: Arm 2: Dapagliflozin+Metformin XR+Placebo vs Arm 3: Saxagliptin+Dapagliflozin+Metformin XR; LOCF; Test type: Superiority or Other; p = 0.0639, ANCOVA — Each secondary endpoint was tested at alpha=0.05; significance testing stops at the endpoint where p-value>0.05; Mean Difference (Final Values) = -9.1, 95% CI 2-sided [-18.8 to 0.5], Standard Error of Mean 4.923

3. Secondary Outcome: Adjusted Mean Change From Baseline in Fasting Plasma Glucose (FPG) at Week 24
Description: Baseline was defined as the last assessment on or prior to the date of the first dose of the double-blind study medication. FPG measurements were obtained at Week 24 in the doubleblind period, including observations prior to rescue.
Time Frame: Baseline (Week 0) and at Week 24
Population: All randomized participants who received study medication and had nonmissing PPG values at baseline and Week 24
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Arm 1: Saxagliptin+Metformin XR+Placebo | Arm 2: Dapagliflozin+Metformin XR+Placebo | Arm 3: Saxagliptin+Dapagliflozin+Metformin XR
Number analyzed (Participants) | 142 | 148 | 155
mg/dL | -14.0 [-19.6 to -8.4] | -31.7 [-37.3 to -26.2] | -37.8 [-43.2 to -32.3]
Statistical Analysis 1: Comparison: Arm 1: Saxagliptin+Metformin XR+Placebo vs Arm 3: Saxagliptin+Dapagliflozin+Metformin XR; Test type: Superiority or Other; Mean Difference (Final Values) = -23.8, 95% CI 2-sided [-31.6 to -15.9], Standard Error of Mean 3.988 — ANCOVA was applied for comparison, but p-value was not reported because at least one prior test in the hierarchical testing procedure yielded p-value>0.05
Statistical Analysis 2: Comparison: Arm 2: Dapagliflozin+Metformin XR+Placebo vs Arm 3: Saxagliptin+Dapagliflozin+Metformin XR; Test type: Superiority or Other; Mean Difference (Final Values) = -6.1, 95% CI 2-sided [-13.8 to 1.7], Standard Error of Mean 3.957 — [estimate comment as in outcome 3, analysis 1]

4. Secondary Outcome: Adjusted Percentage of Participants Achieving a Therapeutic Glycemic Response (Hemoglobin A1c [HbA1C]) <7.0% at Week 24 (Last Observation Carried Forward [LOCF])
Description: Therapeutic glycemic response is defined as HbA1c <7.0%. Data after rescue medication was excluded from this analysis. HbA1c was measured as a percent of hemoglobin.
Time Frame: At Week 24
Population: All randomized participants who received study medication and were not missing baseline and Week 24 (LOCF) values
Measure: Number (95% Confidence Interval); unit: % of Participants
Arm/Group | Arm 1: Saxagliptin+Metformin XR+Placebo | Arm 2: Dapagliflozin+Metformin XR+Placebo | Arm 3: Saxagliptin+Dapagliflozin+Metformin XR
Number analyzed (Participants) | 175 | 173 | 177
% of Participants | 18.3 [13.0 to 23.5] | 22.2 [16.1 to 28.3] | 41.4 [34.5 to 48.2]
Statistical Analysis 1: Comparison: Arm 1: Saxagliptin+Metformin XR+Placebo vs Arm 3: Saxagliptin+Dapagliflozin+Metformin XR; Test type: Superiority or Other; Mean difference in percentages = 23.1, 95% CI 2-sided [14.7 to 31.5], Standard Error of Mean 4.282 — Modified Logistic Regression was applied for comparison, but p-value was not reported because at least one prior test in the hierarchical testing procedure yielded p-value>0.05
Statistical Analysis 2: Comparison: Arm 2: Dapagliflozin+Metformin XR+Placebo vs Arm 3: Saxagliptin+Dapagliflozin+Metformin XR; Test type: Superiority or Other; Mean difference in percentages = 19.1, 95% CI 2-sided [10.1 to 28.1], Standard Error of Mean 4.587 — [estimate comment as in outcome 4, analysis 1]

5. Secondary Outcome: Adjusted Mean Change From Baseline in Body Weight at Week 24
Description: Baseline was defined as the last assessment on or prior to the date of the first dose of the double-blind study medication. Body weight measurements were obtained at Week 24 in the doubleblind period, including observations prior to rescue.
Time Frame: Baseline (Week 0) and at Week 24
Population: All randomized participants who received study medication and had nonmissing body weight values at baseline and Week 24
Measure: Mean (95% Confidence Interval); unit: Body weight Kg
Arm/Group | Arm 1: Saxagliptin+Metformin XR+Placebo | Arm 2: Dapagliflozin+Metformin XR+Placebo | Arm 3: Saxagliptin+Dapagliflozin+Metformin XR
Number analyzed (Participants) | 145 | 152 | 159
Body weight Kg | 0.00 [-0.48 to 0.49] | -2.39 [-2.87 to -1.91] | -2.05 [-2.52 to -1.58]
Statistical Analysis 1: Comparison: Arm 1: Saxagliptin+Metformin XR+Placebo vs Arm 3: Saxagliptin+Dapagliflozin+Metformin XR; Test type: Superiority or Other; Mean Difference (Final Values) = -2.05, 95% CI 2-sided [-2.73 to -1.37], Standard Error of Mean 0.3451 — [estimate comment as in outcome 3, analysis 1]

ADVERSE EVENTS:
Time Frame: 24 weeks
Groups:
- SAXA + MET: Drug: Saxagliptin Tablets, Oral, 5mg , Once daily, 24 weeks Other Names: Onglyza Drug: Metformin XR Tablets, Oral, ≥ 1500mg/≤ 2000mg, Once daily, 24 weeks Other Names: Glucophage XR Drug: Placebo matching with Dapagliflozin Tablets, Oral, 0mg, Once daily, 24 weeks
- DAPA + MET: Drug: Metformin XR Tablets, Oral, ≥ 1500mg/≤ 2000mg, Once daily, 24 weeks Other Names: Glucophage XR Drug: Dapagliflozin Tablets, Oral, 10mg , Once daily, 24 weeks Other Names: BMS512148 Drug: Placebo matching with Saxagliptin Tablets, Oral, 0mg, Once daily, 24 weeks
- SAXA + DAPA + MET: Drug: Saxagliptin Tablets, Oral, 5mg , Once daily, 24 weeks Other Names: Onglyza Drug: Metformin XR Tablets, Oral, ≥ 1500mg/≤ 2000mg, Once daily, 24 weeks Other Names: Glucophage XR Drug: Dapagliflozin Tablets, Oral, 10mg , Once daily, 24 weeks Other Names: BMS512148
Arm/Group | SAXA + MET | DAPA + MET | SAXA + DAPA + MET
Serious Adverse Events (participants affected / at risk) | 6/176 | 2/179 | 2/179
Other Adverse Events (participants affected / at risk) | 0/176 | 0/179 | 0/179
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SAXA + MET (N=176) | DAPA + MET (N=179) | SAXA + DAPA + MET (N=179)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
PANCREATITIS CHRONIC (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
UMBILICAL HERNIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
CHEST PAIN (General disorders) | 1 (1) | 0 (0) | 0 (0)
TOOTH INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
PATELLA FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
GASTRIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less